CLINICAL TRIAL: NCT03571763
Title: The Impact of Anti-thrombosis on Cerebral Microbleeds and Intracranial Hemorrhage in Ischemic Stroke Patients: Prospective, Multi-center, Cohort Study
Brief Title: The Impact of Anti-thrombosis on Cerebral Microbleeds and Intracranial Hemorrhage in Ischemic Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurological department, General Hospital of Shenyang Military Region
Other Study IDs: k(2017)33
Record Dates: First submitted 2018-06-05; First posted 2018-06-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: Cerebral Hemorrhage; anti-thrombosis
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute ischemic stroke patient: acute ischemic stroke patient acute ischemic stroke patient Patient age ≥18 years .Acute ischemic stroke patient confirmed by imaging(SWI sequence) .Time of onset: within 3 months
  Interventions: Other: SWI sequence

INTERVENTIONS:
Other: SWI sequence — Acute ischemic stroke patient confirmed by SWI sequence

SUMMARY:
The purpose of this prospective cohort study is to investigate whether antithrombotic therapy in the secondary prevention of ischemic stroke increases the risk of the emerging CMBs and whether the change is associated with an increased risk of intracranial hemorrhage, providing an imaging evidence for individualized antithrombotic therapy in such patients.

DETAILED DESCRIPTION:
Cerebral microbleeds（CMBs） is a subclinical lesion caused by microvascular disease in the brain, characterized by microleakage of blood. About 30% of ischemic stroke patients, 40% of the healthy people over 80 years old, and 60% of intracranial hemorrhage patients have microbleeds. With the development of imaging technology, clinically more and more patients have found microbleeds in the brain. How these patients are treated with antithrombotic drugs is not yet clear and is in urgent need of evidence. There are only a few prospective cohort studies to determine whether antithrombotic therapy increases the risk of intracranial hemorrhage in ischemic stroke patients with CMBs, but the results are uncertain. More importantly, whether antithrombotic therapy increases the incidence of the emerging CMBs, and whether the change of increased microbleeds is associated with increased intracranial hemorrhage has not been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18 years;
2. Acute ischemic stroke patient confirmed by imaging;
3. Time of onset: within 3 months;
4. Baseline SWI sequence is completed before starting the secondary prevention of ischemic stroke;
5. Baseline SWI sequence must have at least one CMB ;
6. NIHSS≤10

Exclusion Criteria:

1. MRI contraindication;
2. Hemorrhagic transformation after acute Ischemic stroke;
3. Contraindication for antiplatelet or anticoagulation therapy;
4. Severe head trauma or intracranial hemorrhage occurred in the past six months;
5. obvious coagulopathy;
6. Other intracranial lesions associated with (such as tumor, cerebral vascular malformation);
7. other unqualified patients judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ischemic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 1875 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
all cerebral bleeding events | 360 days
  incidence of both cerebral microbleeds and intracranial hemorrhage, determined by MRI

SECONDARY OUTCOMES:
all cerebral bleeding events | 180 days
  incidence of both cerebral microbleeds and intracranial hemorrhage, determined by MRI
proportion of mRS 0-1. | 180、360 days
  the minimum and maximum values of modified Rankin Score (mRS) are 0 and 6, respectively; higher score mean a worse outcome
proportion of cerebral microbleeds | 180 、360 days
  cerebral microbleeds, determined by MRI
proportion of cerebral hemorrhage | 180、360 days
  cerebral hemorrhage, determined by MRI
the occurence of stroke or other vascular events | 180、360 days
the occurence of death due to any cause | 180、360 days

CONTACTS AND LOCATIONS:
Overall Officials: chen huisheng, doctor, Study Director — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China

IPD SHARING:
Plan to Share IPD: No